CLINICAL TRIAL: NCT02397044
Title: Immediate and Early Loading of Hydrothermally Treated, Hydroxyapatite-Coated Dental Implants:a Controlled Randomized Prospective Clinical Study
Brief Title: "Prospective Evaluation of Immediate & Early Loading of Zimmer Hydroxyapatite Coated Dental Implants"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Zimmer Dental (Industry)
Responsible Party: Principal Investigator, David E. Simmons D.D.S., Assistant Professor Department of Periodontics, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: IRB 7438
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Missing Tooth
Keywords: Implants, stability, loading
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Implant loading Immediate: Dental implant surgery with immediate loading
  Interventions: Procedure: Implant surgery
- Implant Loading Early: Dental implant surgery with delayed loading
  Interventions: Procedure: Implant surgery

INTERVENTIONS:
Procedure: Implant surgery — Compare surgical protocols

SUMMARY:
The purpose of this study is to compare the success rates of two surgical protocols. One protocol will have the implants placed at the time of tooth extraction and placed into function. The other protocol will have the implants placed into healed extraction sites and placed into function.

DETAILED DESCRIPTION:
Forty-eight patients (22 men, 26 women) were enrolled in the study and received 48 implants. The population was divided into 2 groups: Group A implants (n=23) were loaded immediately on the day of surgery and Group B implants (n=19) were loaded 3 weeks after surgery. Cone Beam Computed Tomography (CBCT) scans were taken preoperatively to aid in treatment planning. Bone density was evaluated on CBCT scans in Hounsfield units (HU) and by tactile feedback during surgery. Insertion torque was recorded at time of implant placement. Resonance frequency analysis, performed on the day of surgery, at the time of loading, and at 6, 12 and 24 months, was used to record implant stability according to the unit's Implant Stability Quotient (Osstell ISQ). Standardized radiographs were taken at time of implant placement and at 6, 12 and 24 months to measure crestal bone stability. Bone level changes were measured by software (Image J, available online at: http://rsbweb.nih.gov/ij/download.html; last accessed 28 August 2014).

ELIGIBILITY:
Inclusion Criteria:

1. May be either male or female
2. Must be at least 18 years of age
3. Must be of sufficiently good health to undergo routine dental treatment. including the surgical procedures associated with placement of dental implants.
4. Must be partially edentulous requiring single dental implants in their maxilla or mandible
5. Must have sufficient amount of native bone or healed bone grafted sites (by socket grafting, maxillary sinus augmentation and ridge augmentation).
6. Must not have any active infection
7. Must have adequate bone height for at least a 10mm long dental implant
8. Must be physically, emotionally and financially able to undergo the surgical procedure planned
9. Must be adequately compliant

   -

Exclusion Criteria:

1. Have any requirements for antibiotic premedication for infective endocarditis, artificial joints or any other condition
2. Have uncontrolled hypertension
3. Have uncontrolled diabetes
4. Are serological HIV positive
5. Have a history of significant heart, stomach, liver, kidney, blood, immune system or other organ impairment or systemic disease that would prevent their undergoing the proposed treatment
6. Smoke cigarettes or use other tobacco products
7. Have taken any investigational drugs anytime in the previous month
8. Have dental conditions likely to require treatment, necessitating exit from the study such as deep cavities, abscesses, or moderate-severe gum disease
9. Have had radiation therapy to the head and neck
10. Are unwilling or unable to sign the informed consent
11. Don't demonstrate willingness to return for a required number of visits
12. Need an immediate dental implant placement following tooth extraction

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers over the age of 18 needing a tooth replacement.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint Measurement: Implant survival | 6 months
  The primary endpoint for this protocol is implant survival.
Secondary Endpoint Measurements: Crestal Bone Loss, ISQ | 1 year
  Implant survival
  * Crestal Bone Loss will be determined radiographically and will be defined as having occurred when greater than 1.5 mm of bone loss is evident. This endpoint will be summarized for the subgroups of the study population which are formed by stratifying on implant diameter, implant length, implant location and patient age. Rates of crestal bone loss will be computed at one year.
  * ISQ will be measured at the time of implant placement, at 5 months and at one year post implant placement. Insertion torque will be measured at time of placement only.

CONTACTS AND LOCATIONS:
Overall Officials: David E Simmons, D.D.S., Principal Investigator — LSU Helath Sciences Center